CLINICAL TRIAL: NCT00080353
Title: Phase II Study in Metastatic Melanoma Using Lymphocytes Reactive With the gp100 Antigen and Immunization Using a Recombinant rF-gp100P209 Virus Encoding a gp100 Peptide Following a Nonmyeloablative Lymphocyte Depleting Regimen
Brief Title: Vaccine Treatment in Combination With IL-2 and Treated Lymphocytes for Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040152; 04-C-0152; NCT00084500 (obsolete NCT alias)
Record Dates: First submitted 2004-03-27; First posted 2004-03-29 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma
Keywords: Complete Tumor Regression; Cell Survival; Chemotherapy Preparative Regimen; IL-2; Toxicity; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; PMEL protein, human; Muromonab-CD3; montanide ISA 51

INTERVENTIONS:
Drug: IL-2
Drug: gp100:209-217
Drug: OKT3
Drug: rF-go 100P209
Drug: Montanide ISA 51

SUMMARY:
This study will examine the effectiveness of treating advanced melanoma with special tumor-fighting cells taken from the patient's blood or tumor and grown in the laboratory. The cells are given along with infusions of a growth factor-like substance called interleukin-2 (IL-2) and an experimental vaccine called fowlpox gp100. This vaccine consists of a peptide (part of a protein) called gp100 that is often found in melanoma tumors and chicken virus (fowlpox) that has been altered so that it cannot produce illness in humans.

Patients 16 years of age and older with melanoma that has spread beyond the original site and that does not respond to standard treatment may be eligible for this study. Candidates are screened with a medical history and physical examination, chest x-ray, electrocardiogram, blood and urine tests, and x-rays and scans to the evaluate the extent and size of the tumor. Because the experimental preparation is based on tissue type, only patients with tissue type HLA-A*0201 may participate. Tissue type is determined by a blood test.

Participants undergo the following procedures:

* Leukapheresis, a procedure for collecting lymphocytes (white blood cells): Using this procedure, special cells with good tumor-fighting ability are selected and removed for later re-infusion into the patient. To collect the cells, blood is withdrawn through a needle in an arm vein and directed through a catheter into a cell-separating machine. The lymphocytes are removed and the rest of the blood is returned to the body through the same needle. Alternatively, lymphocytes may also be collected from biopsied tumor tissue, obtained either with a needle or by a small cut in the tumor.
* G-CSF injections: This growth factor is injected under the skin every day for 5 days to stimulate white blood cell production.
* Catheter placement: Upon admission to the Clinical Center for treatment, the patient has a catheter (plastic tube) placed in a vein in the neck or arm for giving chemotherapy and other medicines, for infusing the lymphocytes, and for collecting blood samples.
* Leukapheresis: Repeated in the hospital to collect and store blood that may be needed in the rare event that the patient's blood components do not recover after chemotherapy.
* Chemotherapy: A week before the lymphocyte infusion, patients receive a 1-hour infusion of cyclophosphamide for 2 days and then a 15- to 30-minute infusion of fludarabine for 5 days to suppress the immune system and thereby prevent rejection of the infused lymphocytes.
* Vaccine and lymphocyte delivery: The vaccine is injected through the catheter, followed by a 30-minute infusion of the lymphocytes.
* IL-2 and G-CSF: Patients receive IL-2 infusions every 8 hours for up to 5 days after the cell infusion to help keep the cells alive, and G-CSF injections under the skin every day after the cell infusion until white cells increase to a sufficient number. The entire hospital stay is usually 12 to 16 days.

About 4 weeks after the lymphocyte infusion, patients are re-admitted to the hospital for about 10 days for a second vaccine injection and course of IL-2 infusions. Between 2 and 4 weeks after completing the full treatment regimen, patients return to NIH for evaluation. Those whose tumors have shrunk or remained stable may repeat the entire treatment regimen two times. Those whose tumors continued to grow may be re-treated with infusion of lymphocytes through an artery instead of a vein if their tumors receive blood from a major artery. If this is not feasible, or if it is tried without success, the patients will be taken off the study.

DETAILED DESCRIPTION:
Background:

Recent clinical studies in the Surgery Branch have demonstrated clinical responses in patients undergoing adoptive transfer of autologous tumor reactive lymphocytes following a non-myeloablative immunosuppressive chemotherapy regimen. Additional studies in the Surgery Branch using immunization with recombinant fowlpox virus after cell transfer in the immunosuppressed host have provided strong evidence to suggest that the adoptive transfer of lymphocytes in our clinical protocols in patients with melanoma will be substantially improved by the simultaneous administration of recombinant fowlpox virus.

Objectives:

The primary objective will be to determine whether gp100 reactive lymphocytes infused in conjunction with immunization with rf-gp100P209 and administration of high dose or low dose IL-2 may result in complete clinical tumor regression in patients with metastatic melanoma receiving a nonmyeloablative but lymphoid depleting preparative regimen. Secondary objectives will be to determine the survival in patients, of infused cells following this regimen, and to determine the safety of this regimen.

Eligibility:

Patients who are HLA-A201+ must be greater than or equal to 16 years of age and have measurable metastatic melanoma that is refractory to standard therapy. Safety laboratory values must be within defined parameters. More than four weeks must have elapsed since any prior systemic therapy. Patients must be eligible to receive IL-2 and may not have cardiac, pulmonary or other major medical illnesses. Patients may not be allergic to eggs or hypersensitivity to any agents used in this trial, must not require concomitant therapy with steroids.

Design:

Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine and then will be treated by the adoptive transfer of lymphocytes reactive with the gp100:209-217 melanoma antigen, immunization with intravenous fowlpox virus rF-gp100P209, and the administration of high dose or low dose IL-2. Approximately 28 days after the cell infusion, patients receiving high dose IL-2 will receive a second intravenous fowlpox virus rf-gp100P209 followed by administration of high dose IL-2. A complete evaluation of evaluable lesions will be conducted 6-8 weeks after cell infusion. Patients receiving low dose IL-2 will receive a second intravenous fowlpox virus rf-gp100P209 after the 6 weeks of injections and one week of rest followed by repeat administration of the six week cycle of low dose IL-2. A complete evaluation of evaluable lesions will be conducted 3 weeks after the last dose of low dose IL-2. For each of the two cohorts, a small optimal Phase II design will be used and will target 15% (p1=0.15) as a goal for complete response as opposed essentially zero probability normally associated with patients who relapse after high dose IL-2 alone (p0=0.02 will be used). Initially, 16 patients will be enrolled and evaluated in each cohort; if at least 1 of the first 16 patients has a complete response, then accrual to 29 patients will take place. It is expected that it will require 2-3 years to accrue all 58 patients to this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have gp100 reactive cells obtained and evaluated while participating in the Surgery Branch protocol, 'Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols' or on another IRB approved Surgery Branch adoptive cell therapy study, i.e. 99-C-0158 or 03-C-0162.

Patients must be greater than or equal to 16 years of age and must have measurable metastatic melanoma that is refractory to standard therapy, or has relapsed after standard therapy, including high dose IL-2 therapy.

Patients must be HLA-A*0201 positive.

Patients of both genders must be willing to practice birth control during treatment and for four months after receiving the preparative regimen.

Clinical performance status of ECOG 0, 1.

Absolute neutrophil count greater than 1000/mm3 without support of filgrastim.

Platelet count greater than 100,000/mm3.

Hemoglobin greater than 8.0 g/dl (can be corrected with transfusion).

Serum ALT/AST less than three times the upper limit of normal.

Serum creatinine less than or equal to 2.0 mg/dl.

Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

Must be willing to sign a durable power of attorney.

Patients must be able to understand and sign the Informed Consent document.

Patients with resected brain metastases will be eligible.

Patients who are to receive high dose IL-2 and who are 50 years old or greater must have a normal stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) with an LVEF greater than 45 percent.

Patients who are to receive high dose IL-2 who have history of EKG abnormalities, symptoms of cardiac ischemia or arrythmias must have a normal stress cardiac test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) with an LVEF greater than 45 percent.

Patients who are to receive high dose IL-2 who have a prolonged history of cigarette smoking or symptoms of respiratory dysfunction must have a normal pulmonary function test as evidenced by a FEV(1) greater than 60 percent predicted.

CELL INFUSION EXCLUSION CRITERIA:

Less than four weeks has elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, or less than six weeks since prior nitrosurea therapy. All patients' toxicities must have recovered to a grade 1 or less or as specified in the above eligibility criteria. Patients may have undergone minor surgical procedures with the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in section 2.1.1.

Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.

Life expectancy of less than three months.

Systemic steroid therapy required.

Any active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.

Any form of primary or secondary immunodeficiency. Must have recovered immune competence after chemotherapy or radiation therapy as evidenced by normal lymphocyte counts greater than 500 (grade 3 toxicity), normal ANC greater than 1000/mm3 and absence of opportunistic infections. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)

Seropositive for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)

Patients with hepatitis B or hepatitis C will be excluded.

Seronegative for Epstein-Barr virus (EBV).

Allergy to eggs or any known hypersensitivity to any known agents on this trial.

Patients who are not willing to complete a DPA will be excluded.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA, Yannelli JR, Yang JC, Topalian SL, Schwartzentruber DJ, Weber JS, Parkinson DR, Seipp CA, Einhorn JH, White DE. Treatment of patients with metastatic melanoma with autologous tumor-infiltrating lymphocytes and interleukin 2. J Natl Cancer Inst. 1994 Aug 3;86(15):1159-66. doi: 10.1093/jnci/86.15.1159. PMID 8028037
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2004-C-0152.html